CLINICAL TRIAL: NCT02315482
Title: Effect of Pneumoperitoneum and Steep Trendelenburg on Autonomic Nervous System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ASST Fatebenefratelli Sacco (Other)
Collaborators: Andrea Marchi (Unknown); Ferdinando Raimondi (Unknown); Alberto Porta (Unknown); Stefano Guzzetti (Unknown); Tommaso Fossali (Other)
Responsible Party: Principal Investigator, Riccardo Colombo, Autonomic activity during laparoscopic prostatectomy, ASST Fatebenefratelli Sacco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Prostate2
Record Dates: First submitted 2014-11-24; First posted 2014-12-12 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Autonomic Nervous System
Keywords: autonomic nervous system; heart rate variability; prostatectomy; steep trendelenburg; pneumoperitoneum; Intervention Affecting Autonomic Nervous System
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): after induction of general anesthesia (i) a pneumoperitoneum is induced then (ii) patient is placed in steep trendelenburg position at 25 degrees head down
  Interventions: Procedure: pneumoperitoneum insufflation and steep trendelenburg
- Group B (Experimental): after induction of general anesthesia (i) the patient is placed in steep trendelenburg position at 25 degrees head down then (ii) a pneumoperitoneum is induced
  Interventions: Procedure: pneumoperitoneum insufflation and steep trendelenburg

INTERVENTIONS:
Procedure: pneumoperitoneum insufflation and steep trendelenburg — the sequence of pneumoperitoneum insufflation and steep trendelenburg positioning is randomized

SUMMARY:
The purpose of this study is to assess the different effects of pneumoperitoneum and steep trendelenburg position on autonomic nervous system modulation during laparoscopic prostatectomy

DETAILED DESCRIPTION:
Laparoscopic radical prostatectomy is becoming a widely used surgical procedure because it carries some important advantages over open prostatectomy. This surgical technique requires positioning the patient at 25-40 degree head-down position (steep trendelenburg) for a prolonged time in association with pneumoperitoneum at 12-15 mmHg. The postural change from supine to head down position causes a hydrostatic fluid shift towards the head and the thorax, thus increasing venous return and stimulating the cardiopulmonary baroreceptors. Moreover, there are reports of severe bradycardia and cardiac arrest following pneumoperitoneum in association with steep trendelenburg. A vagal hypertone induced by the combination of these two factors, or sympathetic hyperactivity elicited by pneumoperitoneum insufflation have been alternatively advocated as a cause of such hemodynamic changes. However these speculations are little more than a narrative role because any evidence based demonstration is never been provided.

The aim of this study is to measure the variations of autonomic nervous system modulation induced by steep trendelenburg position at 25 degrees and pneumoperitoneum during laparoscopic radical prostatectomy.

Methods Patients are randomized into two groups. Group A: after induction of general anesthesia, in supine position a pneumoperitoneum is induced with carbon dioxide insufflation through a surgical inserted trocar into the abdominal cavity, then patients are positioned in steep trendelenburg at 25 degrees head down. Group B: after induction of general anesthesia, patients are positioned in steep trendelenburg position at 25 degrees head down, then a pneumoperitoneum is induced with carbon dioxide insufflation through a surgical inserted trocar into the abdominal cavity.

Autonomic nervous system modulation is assessed at four main time: (i) T1 baseline (before the induction of general anesthesia); (ii) T2, 5 min after the induction of general anesthesia, (iii) T3, pneumoperitoneum insufflation (Group A) or steep trendelenburg (Group B); (iv) T4, steep trendelenburg (Group A) or pneumoperitoneum insufflation (Group B).

Autonomic nervous system modulation is studied non invasively by means of heart rate variability (HRV) analysis through both linear and non linear methods. Beat-to-beat intervals are computed detecting the QRS complex on the electrocardiogram and locating the R-apex using parabolic interpolation. The maximum arterial pressure within each R-to-R interval is taken as systolic arterial pressure (SAP). Sequences of 300 values are randomly selected inside each experimental condition.

Linear HRV analysis The power spectrum is estimated according to a univariate parametric approach fitting the series to an autoregressive model. Autoregressive spectral density is factorized into components each of them characterized by a central frequency. A spectral component is labeled as LF if its central frequency is between 0.04 and 0.15 Hz, while it is classified as HF if its central frequency is between 0.15 and 0.4 Hz. The HF power of R-to-R series is utilized as a marker of vagal modulation directed to the heart , while the LF power of SAP series is utilized as a marker of sympathetic modulation directed to vessels. The ratio of the LF power to the HF power assessed from R-to-R series is taken as an indicator sympatho-vagal balance directed to the heart. Baroreflex control in the low frequencies is computed as the square root of the ratio of LF(RR) to LF(SAP). Similarly baroreflex control in the high frequencies is defined as the square root of the ratio of HF(RR) to HF(SAP).

Non linear HRV analysis The symbolic analysis is conducted on the same sequences of 300 consecutive heart beats used for the autoregressive analysis. The whole range of the R-to-R interval into each series is uniformly divided in 6 slices (symbols) and pattern of 3 consecutive heart beat intervals are considered. Thus each sequence of 300 heart beats has its own R-to-R range and 298 consecutive triplets of symbols. The Shannon entropy of the distribution of the patterns is calculated to provide a quantification of the complexity of the pattern distribution. All triplets of symbols are grouped into 3 possible patterns of variation: (i) no variation (0V, all 3 symbols were equal), (ii) 1 variation (1V, 2 consequent symbols were equal and the remaining symbol was different), (iii) patterns with at least 2 variations (2V, all symbols were different from the previous one). Previously, the percentage of 0V patterns was found to increase (and 2V decrease) in response to sympathetic stimuli, whereas 2V patterns increased (and 0V decreased) in response to vagal stimuli.

Researcher who analyzes the HRV is blinded to the patient's group assignment.

Management of general anesthesia is standardized as follows:

induction with propofol 1.5-2 mg/kg, Remifentanil Target Controlled Infusion (TCI) Ce 4 ng/ml , neuromuscular blockade with cisatracurium 0.2 mg/kg.

Maintenance: Sevoflurane 0.6-1.5 minimum alveolar concentration (State Entropy target: 40-60); Remifentanil TCI (range Ce 3-15 ng/ml).

mechanical ventilation at respiratory rate ≥14 breaths/min, with tidal volume adjusted to maintain end-tidal carbon dioxide at 32-38 mmHg, and airway plateau pressure <32 cmH2O.

Sample size:

to detect a difference in mean HF(RR) between groups at the trendelenburg positioning of 40 msec^2 with a standard deviation of 50 msec^2 with a power of 0.80 and type I error of 0.05, 26 patients are needed for each group.

ELIGIBILITY:
Inclusion Criteria:

* males scheduled for elective laparoscopic prostatectomy
* sinus rhythm at electrocardiogram
* ectopic heart beats <5% of all heart beats
* american society of anesthesiologists status 1-3

Exclusion Criteria:

* autonomic dysfunction (documented or suspected)
* adrenal or thyroid dysfunction
* organ dysfunction secondary to diabetes (i.e. nephropathy, retinopathy, neuropathy)
* history of stroke, traumatic spinal injury, heart surgery or major vascular surgery
* intracranial hypertension (documented or suspected)
* hydrocephalus
* New York Heart Association cardiac functional status ≥ IIb
* non sinusal heart rhythm
* ectopic heart beats ≥5% of normal heart beats
* therapy with beta-blockers or beta2-agonists

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
changes of High Frequency and Low Frequency spectral heart rate power induced by pneumoperitoneum and steep trendelenburg | 60 min
  changes of autonomic nervous system activity independently elicited by (i) pneumoperitoneum and (ii) steep trendelenburg position. The High Frequency and Low Frequency spectral power of beat-to-beat heart intervals will be assessed with autoregressive analysis and expressed in msec^2

SECONDARY OUTCOMES:
changes of symbolic patterns induced by pneumoperitoneum and steep trendelenburg | 60 min
  changes of autonomic nervous system activity independently elicited by (i) pneumoperitoneum and (ii) steep trendelenburg position. The autonomic nervous activity will be analyzed by means of symbolic analysis of beat-to-beat heart intervals and expressed as percentage of triplets

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Luigi Sacco Hospital, Milan
  - Istituto Clinico Humanitas, Rozzano

REFERENCES:
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Akselrod S, Gordon D, Ubel FA, Shannon DC, Berger AC, Cohen RJ. Power spectrum analysis of heart rate fluctuation: a quantitative probe of beat-to-beat cardiovascular control. Science. 1981 Jul 10;213(4504):220-2. doi: 10.1126/science.6166045.
- [Background] Charkoudian N, Martin EA, Dinenno FA, Eisenach JH, Dietz NM, Joyner MJ. Influence of increased central venous pressure on baroreflex control of sympathetic activity in humans. Am J Physiol Heart Circ Physiol. 2004 Oct;287(4):H1658-62. doi: 10.1152/ajpheart.00265.2004. Epub 2004 Jun 10. PMID 15191897
- [Background] Deutschman CS, Harris AP, Fleisher LA. Changes in heart rate variability under propofol anesthesia: a possible explanation for propofol-induced bradycardia. Anesth Analg. 1994 Aug;79(2):373-7. doi: 10.1213/00000539-199408000-00031. PMID 7639382
- [Background] Falabella A, Moore-Jeffries E, Sullivan MJ, Nelson R, Lew M. Cardiac function during steep Trendelenburg position and CO2 pneumoperitoneum for robotic-assisted prostatectomy: a trans-oesophageal Doppler probe study. Int J Med Robot. 2007 Dec;3(4):312-5. doi: 10.1002/rcs.165. PMID 18200624
- [Background] Ficarra V, Novara G, Artibani W, Cestari A, Galfano A, Graefen M, Guazzoni G, Guillonneau B, Menon M, Montorsi F, Patel V, Rassweiler J, Van Poppel H. Retropubic, laparoscopic, and robot-assisted radical prostatectomy: a systematic review and cumulative analysis of comparative studies. Eur Urol. 2009 May;55(5):1037-63. doi: 10.1016/j.eururo.2009.01.036. Epub 2009 Jan 25. PMID 19185977
- [Background] Gainsburg DM, Wax D, Reich DL, Carlucci JR, Samadi DB. Intraoperative management of robotic-assisted versus open radical prostatectomy. JSLS. 2010 Jan-Mar;14(1):1-5. doi: 10.4293/108680810X12674612014266. PMID 20529522
- [Background] Harrison MH, Rittenhouse D, Greenleaf JE. Effect of posture on arterial baroreflex control of heart rate in humans. Eur J Appl Physiol Occup Physiol. 1986;55(4):367-73. doi: 10.1007/BF00422735. PMID 3758036
- [Background] Hu JC, Gu X, Lipsitz SR, Barry MJ, D'Amico AV, Weinberg AC, Keating NL. Comparative effectiveness of minimally invasive vs open radical prostatectomy. JAMA. 2009 Oct 14;302(14):1557-64. doi: 10.1001/jama.2009.1451. PMID 19826025
- [Background] Guzzetti S, Borroni E, Garbelli PE, Ceriani E, Della Bella P, Montano N, Cogliati C, Somers VK, Malliani A, Porta A. Symbolic dynamics of heart rate variability: a probe to investigate cardiac autonomic modulation. Circulation. 2005 Jul 26;112(4):465-70. doi: 10.1161/CIRCULATIONAHA.104.518449. Epub 2005 Jul 18. PMID 16027252
- [Background] Montano N, Ruscone TG, Porta A, Lombardi F, Pagani M, Malliani A. Power spectrum analysis of heart rate variability to assess the changes in sympathovagal balance during graded orthostatic tilt. Circulation. 1994 Oct;90(4):1826-31. doi: 10.1161/01.cir.90.4.1826. PMID 7923668